CLINICAL TRIAL: NCT04544475
Title: A Randomized, Single Center Pilot Study Comparing Hyaluronic Acid to Vaginal Estrogen for Treatment of Genitourinary Syndrome of Menopause
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: JDS Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-01922
Record Dates: First submitted 2020-09-04; First posted 2020-09-10 (Actual); Results first posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-09

CONDITIONS: Genitourinary Syndrome of Menopause (GSM)
MeSH Terms: interventions — Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Investigational (Experimental)
  Interventions: Device: Revaree
- Standard of Care (Active Comparator)
  Interventions: Drug: Estrace

INTERVENTIONS:
Device: Revaree — Hyaluronic Acid Vaginal Insert (Revaree). A 2g vaginal insert that contains 5mg of HLA sodium salt and a base of semi-synthetic glycerides. It is an insert that does not require an applicator and should be placed in the vagina while laying down twice weekly.
  Other Names: HLA Vaginal Insert
  Arms: Investigational
Drug: Estrace — Vaginal estrogen cream, estradiol: 100mcg
  Other Names: Vaginal estrogen cream
  Arms: Standard of Care

SUMMARY:
Non-hormonal alternatives for the treatment of genitourinary syndrome of menopause (GSM) are needed. In this proposed trial, patients who are diagnosed with GSM will be randomized to receive either a hyaluronic acid (HLA) vaginal insert or vaginal estrogen topical cream for 12 weeks. There will be a baseline visit and an 12 week follow up visit, at which points the patient will undergo a detailed history and physical examination including a pelvic exam, vaginal pH sampling, vaginal cell sample for microscopic analysis, and will fill out a vulvovaginal symptom questionnaire (VSQ). These study arms will be analyzed to assess the efficacy of HLA as compared to the gold standard of vaginal estrogen to treat GSM symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal status as defined by amenorrhea for >12 months or history of bilateral salpingo-oophrectomy or if the patient has had a hysterectomy and menopausal symptoms for >1 year or FSH > 40
2. Symptoms of GSM
3. Negative Pap smear as per ASCCP guidelines
4. Capable of giving informed consent
5. Ambulatory
6. Capable and willing to follow all study-relation procedures

Exclusion Criteria:

1. Use of any HRT (systemic or local) or raloxifene within six weeks of proposed start date
2. History of estrogen-sensitive tumor
3. Undiagnosed vaginal bleeding in the past 12 months
4. History of thromboembolic event
5. Currently have or have had liver problem
6. Bleeding disorder
7. Impaired mental status
8. Prior pelvic irradiation
9. Active vaginal infection
10. Any medical reason the investigator deems incompatible with treatment with vaginal estrogen

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 49 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lila Nachtigall, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be become available beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data upon reasonable request. Requests should be directed to Surbhi.agrawal@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Agrawal S, LaPier Z, Nagpal S, Oot A, Friedman S, Hade EM, Nachtigall L, Brucker BM, Escobar C. A randomized, pilot trial comparing vaginal hyaluronic acid to vaginal estrogen for the treatment of genitourinary syndrome of menopause. Menopause. 2024 Sep 1;31(9):750-755. doi: 10.1097/GME.0000000000002390. Epub 2024 Jul 20. PMID 39042017

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Investigational | Standard of Care
Started | 23 | 26
Completed | 22 | 23
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Investigational | Standard of Care | Total
Number analyzed (Participants) | 23 | 26 | 49
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [57 to 65] | 59.5 [55 to 68] | 59.75 [55 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 26 | 49
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 19 | 22 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 13 | 20 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 23 | 26 | 49

OUTCOME MEASURES:

1. Primary Outcome: Change in VSQ Score
Description: The VSQ (Vulvovaginal Symptoms Questionnaire) is a 21-question survey developed in 2012 that specifically asks about GSM symptoms, their emotional impact, sexual impact, and life impact. Each question is scored from 0 (free of discomfort) to 3 (severe discomfort) The total score ranges from 0 (symptom-free in all areas) to 63 (severe discomfort in all areas) - the higher the score, the more severe the discomfort.
Time Frame: Baseline, Week 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Investigational | Standard of Care
Number analyzed (Participants) | 22 | 23
score on a scale | -3.3 [-5.5 to -1.1] | -3.7 [-6 to -1.3]

2. Secondary Outcome: Change in VMI
Description: VMI (Vaginal Maturation Index) is the microscopic analysis of vaginal tissue that assigns the percentage to the amount of squamous cells visualized. Only the % of squamous cells will be reported in this study since that is most closely correlated with hormonal influence on the vaginal tissue. Vaginal tissue sample will be obtained via scraping for VMI.
Time Frame: Baseline, Week 12
Measure: Mean (95% Confidence Interval); unit: Percentage of squamous cells
Arm/Group | Investigational | Standard of Care
Number analyzed (Participants) | 22 | 23
Percentage of squamous cells | 4.4 [-2.7 to 11.5] | 38.4 [27.6 to 49.2]

3. Secondary Outcome: Change in Vaginal pH
Description: Pelvic samples will be collected to test vaginal pH.
Time Frame: Baseline, Week 12
Measure: Mean (95% Confidence Interval); unit: pH units
Arm/Group | Investigational | Standard of Care
Number analyzed (Participants) | 22 | 23
pH units | -0.2 [-0.3 to -0.1] | -0.3 [-0.4 to -0.1]

4. Secondary Outcome: Change in VAS Score - Dyspareunia
Description: VAS (Visual Analog Scale) score will be reported for dyspareunia. VAS is a visual scale attempting to capture the intensity of a symptom. For each symptom, the score ranges from 0-10. The higher the score, the more severe the symptom. Each symptom will be reported separately.
Time Frame: Baseline, Week 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Investigational | Standard of Care
Number analyzed (Participants) | 22 | 23
score on a scale | -3 [-4.4 to -1.5] | -3.6 [-5.1 to -2.1]

ADVERSE EVENTS:
Time Frame: 12 Weeks
Description: Self-reporting by participants at any point during study or at follow up visit when asked
Arm/Group | Investigational | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/22 | 1/23
Other Adverse Events (participants affected / at risk) | 8/22 | 8/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Investigational (N=22) | Standard of Care (N=23)
Seizure/syncope (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Investigational (N=22) | Standard of Care (N=23)
Urinary Tract Infection (Infections and infestations) | 0 | 1
Vulvovaginal candidasis (Infections and infestations) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Abdominal cramping (Gastrointestinal disorders) | 0 | 1
Tingling in finger (Nervous system disorders) | 0 | 1
Weight gain (Metabolism and nutrition disorders) | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 1 | 1
Vaginal odor (Reproductive system and breast disorders) | 0 | 1
Vaginal discomfort (Reproductive system and breast disorders) | 0 | 1
Vaginal burning sensation (Reproductive system and breast disorders) | 2 | 0
Vaginal irritation (Reproductive system and breast disorders) | 1 | 0
Vulvar itching (Reproductive system and breast disorders) | 1 | 0
Worsening of preexisting condition (Reproductive system and breast disorders) | 1 | 0
Pelvic heaviness (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT04544475/Prot_SAP_000.pdf